CLINICAL TRIAL: NCT03385707
Title: Hypoglycemia and the Gut Microbiome
Status: Active, not recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-28
Record Dates: First submitted 2017-12-07; First posted 2017-12-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypoglycemia
Keywords: Post-bariatric hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or saliva samples are being collected for future genotyping to identify genetic factors linked to risk of hypoglycemia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CGM and Microbiota: Participants will wear a Dexcom continuous glucose monitor (CGM) and activity monitor for two weeks. They will not be aware of sensor glucose values. A stool sample will be collected. The investigators will evaluate relationships between patterns of postprandial glycemia, recorded by CGM, food intake, and microbiome composition.

SUMMARY:
This study is designed to evaluate individuals who are currently experiencing symptoms of hypoglycemia, in order to discern correlations between microbiome composition and patterns of postprandial glycemia.

DETAILED DESCRIPTION:
Recent studies have shown that analysis of the gastrointestinal microbiome can be used to predict glycemic response to dietary intake. Specifically, integrative analysis of dietary consumption, anthropometrics, physical activity and gut microbiota composition can be used to predict postprandial glycemic excursions. The investigators hypothesize that individualized assessment of glycemic responses to food, together with analysis of the gut microbiome, will allow the design of a personalized dietary approach to minimize glycemic excursions for patients with post-bariatric and other forms of largely postprandial hypoglycemia. Identification of factors predictive of glycemic excursions and subsequent hypoglycemia may ultimately allow individuals to tailor their diet towards foods which would not induce hypersecretion of insulin and subsequent hypoglycemia.

ELIGIBILITY:
Inclusion Criteria

1. Males or females diagnosed with ongoing post-bariatric, post-gastric surgery or other forms of postprandial hypoglycemia with prior episodes of neuroglycopenia
2. Age 18-65 years of age, inclusive, at screening.
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria

1. Documented hypoglycemia occurring in the fasting state (> 12 hours fast);
2. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
3. Hepatic disease, including serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
4. Congestive heart failure, New York Heart Association (NYHA) class II, III or IV;
5. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use.
6. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia
7. Concurrent administration of β-blocker therapy;
8. History of a cerebrovascular accident;
9. Seizure disorder (other than with suspect or documented hypoglycemia);
10. Active treatment with any diabetes medications except for acarbose;
11. Active treatment with octreotide or diazoxide;
12. Active malignancy, except basal cell or squamous cell skin cancers;
13. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
14. Known insulinoma;
15. Major surgical operation within 30 days prior to screening;
16. Hematocrit < 33%;
17. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
18. Blood donation (1 pint of whole blood) within the past 2 months;
19. Active alcohol abuse or substance abuse;
20. Current administration of oral or parenteral corticosteroids;
21. Pregnancy and/ or lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intrauterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
22. Use of an investigational drug within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experience hypoglycemia after bariatric or other upper gastrointestinal surgery or those with reactive hypoglycemia in the absence of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of cumulative duration of hypoglycemia | 2 weeks
  Duration of hypoglycemia will be assessed by: (1) the number of minutes per day with hypoglycemia, defined as sensor glucose <70 mg/dl, and (2) the number of minutes per day of severe hypoglycemia, defined as sensor glucose <55 mg/dl. Data will be captured for the entire 24 hour period as well as day and night subsets.

SECONDARY OUTCOMES:
Analysis of frequency of glycemic excursions | 2 weeks
  Hypoglycemia frequency will be assessed by: (1) number of episodes of hypoglycemia, both moderate (55-70 mg/dl) and severe (<55 mg/dl), (2) number of episodes requiring assistance, and (4) number of episodes of hyperglycemia (>180 mg/dl). All data will be averaged and reported as episodes per day.
Impact of activity on glycemic patterns in post-bariatric hypoglycemia | 2 weeks
  Activity measures (total step number per day) will be analyzed to determine relationship to changes in sensor glucose levels. Data will be integrated to determine relationships between glycemic patterns, diet, and microbiome.
Impact of diet on glycemic patterns in post-bariatric hypoglycemia | 2 weeks
  Dietary information will be transcribed and recorded from participants' food diaries. Data will be integrated to determine relationships between glycemic patterns, diet, and microbiome.
Analysis of microbiome in individuals with post-bariatric hypoglycemia | 2 weeks
  Stool samples will be analyzed to determine microbiome community by 18S sequencing. Data will be integrated to determine relationships between glycemic patterns, diet, and microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patti ME, Goldfine AB. The rollercoaster of post-bariatric hypoglycaemia. Lancet Diabetes Endocrinol. 2016 Feb;4(2):94-6. doi: 10.1016/S2213-8587(15)00460-X. Epub 2015 Dec 15. No abstract available. PMID 26701701
- [Background] Mulla CM, Middelbeek RJW, Patti ME. Mechanisms of weight loss and improved metabolism following bariatric surgery. Ann N Y Acad Sci. 2018 Jan;1411(1):53-64. doi: 10.1111/nyas.13409. Epub 2017 Sep 3. PMID 28868615
- [Background] Suhl E, Anderson-Haynes SE, Mulla C, Patti ME. Medical nutrition therapy for post-bariatric hypoglycemia: practical insights. Surg Obes Relat Dis. 2017 May;13(5):888-896. doi: 10.1016/j.soard.2017.01.025. Epub 2017 Jan 16. PMID 28392017